CLINICAL TRIAL: NCT05021523
Title: Heat Therapy to Prevent Deconditioning During Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspetar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: F202007002
Record Dates: First submitted 2021-06-30; First posted 2021-08-25 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hot Weather; Adverse Effect; Immobilization, Tonic
MeSH Terms: conditions — Immobility Response, Tonic | interventions — Immobilization

STUDY DESIGN:
Intervention Model Description: Repeated measure design (pre/post intervention) with an intervention group and a sham group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEAT group (Experimental): Participants are doing passive and active heat exposures
  Interventions: Other: Hot ambient conditions exposures; Other: Immobilization
- CON group (Sham Comparator): Participants are doing sham altitude exposures
  Interventions: Other: Immobilization

INTERVENTIONS:
Other: Hot ambient conditions exposures — Participants rest or exercise for 40min to 1h daily in hot ambient conditions
  Arms: HEAT group
Other: Immobilization — Participants are wearing a walking boot (with crutches) for 2 weeks

SUMMARY:
Animal models suggest that heat stress increases protein content and facilitates the recovery of atrophied muscle after an immobilization period, or following a chemically induced muscle injury in rats. Thus, a recent study in human have reported that daily heat treatments, applied during 10 days of immobilization, reduced the loss of muscle mass. In addition of protecting muscle mass, repeated heat stress may also help to maintain cardiovascular fitness from the onset of injury through passive exposures in the condition that they sufficiently trigger an increase in body temperature, circulation and sweating. This study will investigate the benefits of using heat therapy to prevent deconditioning during immobilization in human.

DETAILED DESCRIPTION:
1.3 Background information & study rationale Heat is often used as a traditional therapy in many cultures to treat a variety of health conditions. At the level of the skeletal muscle, repeated heat exposures have been reported to increase cell proliferation and muscle protein content in vitro and in animal studies. Rodent studies have further shown that repeated heat exposure may reduce muscle atrophy during immobilization and facilitate the recovery of atrophied muscle after immobilization. The effect of heat therapy might also have numerous benefits in humans. For example, repeated passive heat exposure may improve quality of life in different populations, improve cardiovascular health, and is associated with a lower risk of fatal cardiovascular disease and all-cause mortality. Moreover, considering the association between skeletal muscle mass/function and health, two studies demonstrated that 8 to 10 weeks of repeated localized heat therapy induced skeletal muscle adaptations, increasing peak torque.

To our knowledge, the only study conducted in humans reported that daily 2-h of local heat therapy during 10 days of lower limb immobilization was sufficient to reduce vastus lateralis atrophy and maintain mitochondrial function. In rats, a single 60-minute exposure to heat an environmental chamber protects against short-term atrophy of skeletal muscle. In addition, Daily 30-min exposure to similar environmental thermal stress has also been shown to maintain mitochondrial content and oxidative capacity.

The investigators therefore conducted a first study in Aspetar showing that passive heat acclimation (11 days, 1 h per day) improves skeletal muscle contractile function during both normothermic and in the hyperthermic humans. These improvements were verified in measures obtained at rest and during contractions at different intensities ( 10, 25, 50, 75% MVC), as well as in different neuromuscular parameters: an increase in electrically evoked .peak twitch amplitude, an increase in maximal torque production at a similar level of voluntary activation, and an improvement of the relative torque/EMG linear relationship. This infers that passive heat acclimation improves skeletal muscle contractile function in humans, irrespective of thermal state. As such, this highlights a novel passive method to improve muscle function via passive heat exposure that may be used with athletes and patients during a period of musculoskeletal unloading, such as post-surgical immobilization.

1.4 Study goals and objectives The aim of the study is to investigate the benefits of using whole-body heat therapy to prevent deconditioning during immobilization in human 1.5 Study Design and Research Population

1. Scientific justification for the research
2. The type of study Randomized controlled trial
3. Research population or the sampling frame

   1. Total size of subjects across all sites (inside and outside Qatar): 20 volunteers will participate after providing written consent. The participants will be healthy adult males recruited from local institutions (e.g., Aspire, Aspetar).

   2. How was sample size and grouping decided upon: A sample size of 10 participants per group has been calculated using data from a previous work from our group reporting an effect of heat exposure on peak twitch (the main outcome variable for muscle contractility) with a partial eta square of 0.266. G-Power was used to estimate the required sample size with an alpha of 0.05 and a power of 0.9.

   3. Gender: males 4. Age: 18 to 45 yrs 5. Possible inclusion of Vulnerable Population (i.e. Pregnant women, fetuses or neonates, prisoners, children, persons with mental disabilities, economical disadvantages and Fellow employees) N/A 6. Language of participants: All primary language can participate, but participants will have to be able to communicate with the experimenter in English 7. How long will an individual subject participate in the research? 9 weeks 8. How long will it take to enroll all needed subjects? 6 months 9. Power calculation for determining sample size. A sample size of 10 participants per group has been calculated using data from a previous work from our group reporting an effect of heat exposure on peak twitch (the main outcome variable for muscle contractility) with a partial eta square of 0.266. G-Power was used to estimate the required sample size with an alpha of 0.05 and a power of 0.9.
4. Inclusion Criteria Age (18 to 45 yrs); males, Constant level of activity for at least 2 months before the start of the study; Fluent English speaker
5. Exclusion criteria Contraindication to physical activity as per the Par-Q questionnaire; Neural, skin or muscular pathology, contraindication to the MRI
6. Withdrawal criteria The participants will have the freedom to withdraw from the study at any time, without having to give any explanation to the experimenters.
7. Criteria for electively stopping the trial or other research prematurely (if applicable) N/A
8. Procedures and person responsible for recruitment. Potential participants will be originally contacted through the Human subjects Recruiting and Adverting Form (RO-F14, attached). Their will provided with the informed Consent Form (RO-F05, attached) and have the opportunity to speak with the research before to start.
9. Medical screening - who and how. (If applicable) N/A 1.6 Methodology & Project Duration This study will assess the effect of daily heat therapy on skeletal muscle subjected to immobilization. All participants will first undergo 4 weeks of standardized physical conditioning, followed by 2 weeks of limb immobilization and 2 weeks of return to sport (RTS). During immobilization, participants will be assigned, in a counterbalanced fashion, to either HEAT (11 sessions of whole-body passive heat exposure) or CON (sham treatment with the participants being told that they are at an altitude of 3000 m while it remained at 200 m) groups. Throughout return to sport, the HEAT group will perform 5 trainings in the heat whereas the CON group will perform the same training in sham conditions. the tests will be performed the week before the intervention as well as at the end of weeks 4, 6 and 8 of interventions.

Initial training: All participants will be engaged in a structured physical training program for 4 weeks. Each week includes 2 'aerobic' sessions and 3 strength and conditioning sessions.

Immobilization: Prior commencing the immobilization protocol, participants will receive instructions for the use of the therapeutic boots and medical arm crutches. The left ankle of each participant will be immobilized at an angle of 90° for 14 consecutive days. Participants will be instructed to use crutches and not to engage in any weight-bearing activity with the immobilized ankle. They will however, be allowed to ambulate freely throughout the immobilization period. All participants will report to the laboratory six days per week during the immobilization period, during which they will receive either 60 min of whole-body passive heat treatment (i.e., HEAT) or sham treatment (i.e., CON). Heat treatment will be undertaken according to previous methods where participants will assume seated rest in an environmental chamber set at 50°C and 50% relative humidity. The control group will receive sham treatment and will undertake seated rest in altitude room set at 200 m of altitude, 24°C.

Return to sport: Following the immobilization period, participants will be engaged in a structured rehabilitation program for 2 weeks including 5 sessions per week. Three of the sessions will have a general conditioning objective while the 2 others will focus on neuro-muscular training. The HEAT group will perform the three conditioning sessions in an environmental chamber set at 35ºC and 60 % humidity, whilst the CON group will be at 200 m, 22ºC. The remaining two sessions will be performed in standard laboratory conditions.

Data collection procedure

The physical tests will be performed before training (week 0), after training (week 4), after immobilization (week 6) and at return to sports (week 8) (Fig. 1). The biopsy and MRI will be performed after training (week 4), after immobilization (week 6) and at return to sports (week 8) only (Fig. 1). A typical week of testing will include the MRI imaging and physical tests on the Saturday, the questionnaires and proprioception on the Sunday and the biopsy and blood samples on the Monday (i.e., 48h after the physical tests).

Neuromuscular test:

The isometric neuromuscular tests will be conducted on Dynamometric pedal (Captels, St. Mathieu de Treviers, France). The fatigue test will be performed on a isokinetic dynamometer (Biodex System 3, NY, USA).

Electrically evoked twitch: The tibial nerve will be electrically stimulated (voltage400 V, rectangular pulse of 0.2 ms) via a high-voltage stimulator (Digitimer DS7AH; Digitimer, Hertfordshire, UK). through a cathode placed in the popliteal cavity (diameter 9 mm) and an anode placed distally to the patella (5 x 10 cm). The intensity for each participant will be increased progressively (10-mA increment) until a plateau in twitch mechanical response (i.e., peak twitch, PT). The final intensity will be set at 150% of the final plateau, the participant will be stimulated 5 times with 5 s rest between each peak twitch. The twitch evoked will be used to calculate the peak twitch amplitude (Pt), contraction time (CT) and half relaxation time (HRT).

H-Reflex: EMG activity of the soleus and gastrocnemius medialis will be recorded using bipolar surface electrodes. The intensity will be adjusted to obtain maximal soleus H-reflex amplitude. 6 soleus H-reflex responses will be recorded with an interval of 20 sec to avoid post-activation depression. The H-reflex will be normalized by the M-wave recorded during the peak twitch.

Rate of torque development: Participants will receive the instructions to produce 5 maximal contractions as fast as possible. The contractions will be short (~1 s) and interspersed by short rest periods (e.g., 20 s).

Maximal Voluntary contraction: Participants will be required to perform an isometric maximal voluntary contraction (MVC) of the plantar flexors. Participants will be instructed to push as hard as possible against the dynamometric pedal by contracting his plantar flexor muscles. Visual feedback will be given to the participant during the effort, and standardized verbal encouragement. The MVC is reached when a plateau is observed. Double stimulation will be delivered during the plateau of MVC (superimposed twitch), and another double stimulation when the muscle is fully relaxed Immediately after the contraction (potentiated twitch). The ratio between the superimposed and the potentiated twitch will be used to calculate voluntary activation as VA (%) = (1-superimposed twitch/potentiated twitch) x 100. The subject will perform a second MVC of the plantar flexor with at least 1 min rest between each trial, If the peak torque from the second trial is not within 5% of the first, additional trials must be performed. The greatest torque achieved by the subject is taken as the MVC torque. Thereafter, participant will perform a submaximal contraction at 25, 75 and 50 % of the previous MVC to estimate the torque/electromyographic (EMG) relationship.

Fatigue test: Fatigue protocols will be performed on an isokinetic dynamometer with the participants seated with the hip joint at about 80° and knee at 100°. The foot will be placed on the foot adapter with an ankle angle in 10° of plantar flexion and fixed with straps. In order to induce fatigue in the ankle, the participant will perform 30 contractions in concentric mode at 60° s-1 for the plantar flexion and at 90° s-1 for the dorsiflexion (the range of motion is between -25°and 45°). A fatigue resistance index (FRI) will be calculated hinge on the changes in torque over the 30 contractions using the following formula: FRI = (100 x (total PT/Ideal PT)) - 100, where total PT: the sum of PT over 30 contractions, Ideal PT: best PT x 30.

Proprioception testing:

Dynamic balance testing: The Y Balance Test (YBT) will be performed with the participants standing barefoot on the balance test kit™ (a stance platform with three pieces of plastic pipe in the anterior, posteromedial, and posterolateral reach directions). Participants will be asked to reach as far as possible in each direction. Participant will first perform 3 unrecorded practice followed by 3 recorded trial. The outcome measure will be the average of the best 2 properly executed tests for each direction.

Movement discrimination testing: Gibsonian 'obtained' proprioceptive acuity would be assessed at the ankle using a custom-made Active Movement Extend Discrimination Apparatus (AMEDA). The participants will stand with the left leg on a fix support and the right leg on a mobile support. The mobile support will allow the participants to reach 5 different plantar flexion angles. The participants will undergo a total of 50 trials (10 at each angle) and will have to actively recognize the angle allowed.

Questionnaire:

All the questionnaires are hard copy distribution (attached). The Pittsburgh Sleep Quality Index (PSQI) will be used to assess subjective sleep quality over the next month. The PSQI consists of 19 questions measuring seven components: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, the use of sleeping medications, and daytime dysfunction. The total score for the PSQI ranges from 0 to 21, where ''0'' indicates no difficulty and ''21'' indicates severe difficulties in all areas. A PSQI score 5 is considered to indicate poor sleep quality, although a more conservative threshold of 8 may also be used. Based on the above, subjects will be classified as good sleepers (PSQI<=5) and bad sleepers (PSQI>5). In addition, self-reported variables from PSQI component scores provided quantitative data for sleep onset latency (minutes), total sleep time (hours), and sleep efficiency (%; ratio of total sleep time to time in bed for sleep. The questionnaire will be distributed before the begging of the tests. The PSQI is a valid and reliable questionnaire to determine subjective sleep quality. It has a sensitivity of 89.6% and specificity of 86.5% for identifying cases with sleep disorder, using a cut-off score of 5. Validity is further supported by similar differences between groups using PSQI or polysomnographic sleep measures.

The World Health Organization Quality of Life-BREF (WHOQOL-BREF) The instrument is a 26-item self-report inventory, rated on a 5-point Likert-type scale with varying scale response anchors. Two items are intended to measure perceptions of general QOL and health, and the remaining 24 items are designed to measure one of the following four domains of QOL: physical (seven items), psychological (six items), social (three items), and environment (eight items). Only the 24 items used to yield domain scores. The score for each domain varies from zero to 20, zero being considered the worst and 20 the best quality of life.5 For questions one and two the maximum score is 25 points.

The Profile of Mood States Brief questionnaire (POMS Brief questionnaire) consists of 40 adjectival items (e.g., tense, worthless) which was used to measure 7 aspects of mood (tension, depression, anger, vigor, fatigue, esteem-related affect, confusion). Participants rated each item on a five-point answer scale. The score of each mood dimension equals the sum of scores of several particular questions. The total score of abbreviated POMS, called total mood disturbance, is calculated by subtracting the scores of two positive dimensions from the five negative dimensions and adding 100. Therefore, the higher the total score is, the more negative mood one may have Lower extremity functional scale (LEFS): The participants will fill the LEFS to estimate their lower limb function after immobilization and return to sport.

Fitness:

Incremental exercise testing: Each participant performed an incremental cycling test on an electromagnetically braked cycle ergometer (Excalibur, Lode, Groningen, The Netherlands), which will be adjusted to each participant's specifications and with the feet securely strapped on the pedal. The test will commence by 7 min of warm-up (2min at 50 W + 3 min at 1.5 W/kg + 2 min at 50 W) and will thereafter progressively (i.e. ramp) progress by 25 W per minute until volitional exhaustion. Maximal oxygen uptake will be determined by the highest 30 s average upon exercise termination (InnocorTM).

Haemoglobin mass (Hbmass) will be measured using the optimized CO-rebreathing technique. Briefly, participants will be seated for 20-min to allow plasma volume to stabilize. Participants will fully exhale to residual volume into a portable CO sensor (Draeger, Luebeck, Germany) to detect existing levels of CO within the body and baseline fingertip capillary samples (200 μL) will be obtained. Participants will wear a nose-clip and will be connected to a closed spirometer via the mouth piece at the end of a maximal expiration. Participants will be instructed to inhale deeply and hold their breath for 10-s while an individualized bolus (1.2g/kg) of 99.5% medical grade carbon monoxide (CO) is administered via a 150mL syringe. Simultaneously, the valve for a 3L anesthetic bag pre-filled with pure oxygen will be opened. After 10-s participants will be asked to continue normal respiration through the spirometer for 1-min 50-s. During this time, a portable CO analyzer (Draeger Luebeck, Germany) with parts-per-million sensitivity will be held in close proximity to the mouth piece and spirometer to verify that no gas has escaped. After 2-min of re-breathing, the participants will be asked to fully exhale to residual volume or until the anesthetic bag is filled to quantify the amount of CO which was not taken up by the body. Thereafter, the spirometer will be disconnected and the participants will continue to sit quietly. Two minutes later, participants will again fully exhale to residual volume into a portable CO sensor (Draeger, Luebeck, Germany) and combined with the remainder of CO within the spirometer after the test to determine the quantity of CO not taken up by the body. At exactly 7-min after commencement of re-breathing, further fingertip capillary samples (200 μL) will be obtained. All capillary samples will be immediately analyzed in triplicate for percent carboxyhemoglobin (%HbCO) and hematocrit (Hct.) using a spectrophotometer (ABL 90, Radiometer, Denmark). Carbon monoxide leaves the body within 5 hours after the procedure.

Mechanical loading:

Mechanical changes during walking (4 km/h) and running (10 km/h) will be assessed on an instrumented treadmill (HP Cosmos, Germany) with a capacitance-based pressure platform (FDM-THQ, Zebris Medical GmbH, Germany). The treadmill surface will be set at 0° grade for all testing. The capture surface of the Zebris FDM-THQ system is 1.70 × 0.65 m and contains a sensing area of 1.36 × 0.64 m which consists of 10,240 sensors of 0.85 × 0.85 cm each. The sensor threshold will be set at 1 N/cm2 and the measuring range is 1-120 N/cm2. Locomotion at each velocity will be for 60 s, with 60 s rest in-between. Mechanical loading during walking will be assessed prior to training and immobilization, as well as following immobilization and return to sport. Assessment during running will be omitted immediately following immobilization, which otherwise will be undertaken at all other time-points. At each speed, data will be captured for the last 20 s of each minute. Raw data from the Zebris system will be exported, and analyzed for changes in plantar pressure distribution, asymmetry and plantar vertical force.

Biological measures:

Muscle biopsy: Muscle samples will be extracted from the muscle belly of medial gastrocnemius using a disposable, spring-loaded microbiopsy system (MAX-CORE, Bard Biopsy Systems). A 14-gauge biopsy needle will be inserted under local anesthesia (1% xylocaine) after skin incision, and 4 samples, totaling approximately 80 mg will be extracted per biopsy. The tissue samples will be immediately frozen in liquid nitrogen and stored in a -80°C freezer until further analysis. Analyses will include 23 proteins (FGF21, GDF15, Adropin, Irisin, Humanin, SHLPs, MOTS-c, TFAM, Cardiolipin, ND6, P-FOXO3, P-FOXO1, Total FOXO, P-AMPK, Total AMPK, P-4EBP1, Total 4E-BP1, P-P70S6K, Total P70S6K, P-RPS6, Total RPS6, NCAM, PAX7) and 19 mRNAs (UPRmt as measured by ATF5, CHOP, ClpP, HSP10, HSP60; mt DNA as measured by COX1, ND1, ND6, D-loop; Atrogin-1; MuRF-1; HSP 70; PGC-1alpha; Myostatin; Myogenin; MyoD; and 3 housekeeping genes). Participants will be provided with standardized meal for the 2 days preceding the biopsies.

Blood samples: Approximately 16 ml of blood will be drawn from the antecubital vein using standard venipuncture technique. Blood will be drawn into 1 serum (red) and 3 EDTA (purple) vacutainers and will be subsequently centrifuged. The supernatant will be aliquoted to Eppendorf tubes and subsequently stored at -80°C until further analysis. Analyses will include 10 proteins (FGF21, GDF15, Adropin, Irisin, Humanin, SHLP2 or 3, MOTS-c, TFAM, Cardiolipin, ND-6).

Muscle volume:

MRI: T1-weighted Spin Echo Axial Images will be acquired from the knee to the Achilles tendon with the following parameters: FOV 300mm, Image Matrix 240x320, Slice thickness 6mm with 0mm gap, TR/TE = 730/14.

Ultrasound assessment: Muscle thickness, pennation angle, and fascicle length of the Gastrocnemius will be determined from images taken along the longitudinal axis of the muscle belly, by utilizing a two-dimensional, B-mode ultrasound (frequency 12 MHz; depth 8 cm; field of view (FOV) 14×47 mm) (Logiq E, GE Healthcare, IL, USA). The scanning site will be halfway point between the ankle and knee joints.

Ultrasound Tissue Characterization (UTC): UTC imaging utilizes a 5-12MHz ultrasound (US) transducer (SmartProbe 12 L5, Terason 2000, Teratech, USA) fixed in a transverse position into a 12 cm tracking device (UTC Tracker, UTC imaging, Netherlands), allowing the capture and storage of a sequence of transverse images of the tendon at regular intervals of 0.02 cm. The UTC tracking device is maintain in contact with the achilis by the experimenter. The US transducer then moved down the track driven by a motor, from proximal to distal, resulting in a total of 598 sequential transverse images acquired in 45 s. With these scans the UTC algorithm creates a 3D block of the scanned area allowing additional reconstructed coronal and sagittal views.

Anthropometry: Muscle mass and body fat percentages will be assessed by an accredited nutritionist from skinfold thickness (Harpenden, UK). The muscle volume of the leg will be specifically assessed from the leg length and circumferences (i.e. truncated cone methods) along skinfold thickness (Siri 1956, Durnin and Rahaman 1967, Durnin and Womersley 1974, Jones and Pearson 1969).

Core, skin and muscle temperature:

Core temperature will be measured the first and the last day of the intervention period and the RTS period using a e-Celsius® rectal capsules (BodyCap®, Caen, France) . Skin temperatures will be determined using iButton temperature sensors/data loggers (iButtonTM, Maxim Integrated Products, Sunnyvale, CA, USA), secured to the participants' chest, arm, thigh and calf using non-porous adhesive tape. Mean skin temperature will be determined using the following formula: Tsk = (0.3 x Tchest) + (0.3 x Tbicep) + (0.2 x Tthigh) + (0.2 x Tcalf). Muscle temperature will be measured only once (e.g. on the Thursday of week 1) using an indwelling flexible thermistor (MAC flexible probe, Ellab, Hilleroed, Denmark), and inserted via a catheter (16 GA) after local anesthesia of the skin (2 mL of Xylocaine without adrenaline) by a physician.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 yrs old
* Male
* Constant level of activity for at least 2 months before the start of the study
* Fluent English speaker

Exclusion Criteria:

* Contraindication to physical activity as per the Par-Q questionnaire
* Neural pathology
* Muscular pathology
* Contraindication to the MRI

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Change in maximal strength of the plantar flexors from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  Maximal voluntary isometric torque of the right leg (plantar flexors) in N.m
Change in maximal strength of the plantar flexors from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  Maximal voluntary isometric torque of the right leg (plantar flexors) in N.m
Change in muscle volume of the plantar flexors from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  MRI to measure muscle volume
Change in muscle volume of the plantar flexors from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  MRI to measure muscle volume
Change in muscle protein content from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  Muscle biopsy
Change in muscle protein content from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  Muscle biopsy

SECONDARY OUTCOMES:
Change in maximal aerobic capacity from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  VO2max during an incremental test
Change in maximal aerobic capacity from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  VO2max during an incremental test
Change in maximal aerobic power from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  Maximal power reached during an incremental test
Change in maximal aerobic power from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  Maximal power reached during an incremental test
Change in blood volume from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  Blood volumes measured by the CO-rebreathing technique
Change in blood volume from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  Blood volumes measured by the CO-rebreathing technique
Changes in ankle proprioception from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  Active movement extent discrimination assessment (AMEDA) score on the right leg (0 meaning no error, 160 being the maximum total error possible)
Changes in ankle proprioception from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  Active movement extent discrimination assessment (AMEDA) score on the right leg (0 meaning no error, 160 being the maximum total error possible)
Change in voluntary activation of the plantar flexors from baseline to post-immobilization | Baseline (week 4) and week 6 (post immobilization)
  Change in the maximal voluntary activation of the right leg (plantar flexors) in percent estimated by the interpolated twitch technique
Change in voluntary activation of the plantar flexors from baseline to post-retraining | Baseline (week 4) and week 8 (post retraining)
  Change in the maximal voluntary activation of the right leg (plantar flexors) in percent estimated by the interpolated twitch technique

CONTACTS AND LOCATIONS:
Locations (1):
- Aspetar, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No